CLINICAL TRIAL: NCT04555798
Title: The Immunoadsorption Effect of Arterio-venous ECMO in Refractory Septic Shock With ARDS Following Severe Lung Contusion
Brief Title: Effect of Arterio-venous ECMO on Severe Sepsis and ARDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohamed Gaber Allam (Network)
Collaborators: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor-Investigator, Mohamed Gaber Allam, Consultant intensivist, King Abdul Aziz Specialist Hospital
Organization: King Abdul Aziz Specialist Hospital (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ICU-44-20
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Patients With Respiratory Failure and Shocked
MeSH Terms: conditions — Shock | interventions — Meropenem

STUDY DESIGN:
Intervention Model Description: 100 patients from those who showed no improvement after 10 days ventilation and still had respiratory failure and in need of high ventilatory parameters (as mentioned before), fulfilled > 2 parameters on SOFA score as illustrated in table (2), > 6 on CPIS score as illustrated in table (3) and developed circulatory failure (septic shock) with nor-adrenaline infusion and only on high dose of nor-adrenaline included in our study (>5microgram/kg/minute intravenous infusion as circulatory support). Since the parameters of those 100 patients selected are considered indication for arteriovenous extracorporeal membranous (A-V ECMO), so patients randomly allocated in two groups 50 patients in each. Randomization sequence was created using Excel 2007 (Microsoft, Redmond, WA, USA) with a 1:1 allocation using random block sizes of 2 and 4 by an independent doctor. In this way, sequence generation and type of randomization can be expressed at the same time
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Group A (Placebo Comparator): Group A continue on the same conventional way of management as mentioned above with conventional way of ventilation and broad spectrum antibiotics coverage
  Interventions: Drug: Meropenem Injection
- Group B (Active Comparator): group B who connected to (A-VECMO).with venous access from femoral vien and arterial cannulation using the femoral artery
  Interventions: Drug: Meropenem Injection; Device: A-V ECMO

INTERVENTIONS:
Drug: Meropenem Injection — patients of both groups given meropenam 1 gram every 8 hours till we collect the sputum culture
Device: A-V ECMO — Only patients of group B connected to A-V ECMO for two weeks
  Arms: Group B

SUMMARY:
To evaluate and compare the effect of immunoadsorption effect of A-V ECMO on course of sepsis weaning from inotropes, weaning from the ventilator, duration of ICU stays and effect on mortality rate in patients with septic shock and respiratory failure due to ARDS followed severe lung contusion.

DETAILED DESCRIPTION:
100 patients with respiratory failure without improvement after 10 days ventilation due to development of VAP with ARDS, had >2 SOFA score and >6 CPIS score included in two groups 50 patients in each. Only patients of group B put on A-V ECMO while patients of group A continue on traditional way of management. Improvement of ARDS &VAP, weaning from ventilation, duration of ICU stays, improvement of one/all parameters of both SOFA and CPIS scores, morbidity and mortality recorded and compared within 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Those who had an age between 18-65 years old
* patients ventilated for more than 10 days
* with conscious level more than 8/15 on Glasgow Coma Scale

Exclusion Criteria:

pediatric patients below 18 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
number of patients weaned from ventilators | 2 weeks
  who showed improvement in CPIS score
number of patients disharged from ICU | 2 weeks
  who successfully weaned from the ventilator and complete 24 hours observation without symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
only after publishing the work in specific journal